CLINICAL TRIAL: NCT07203638
Title: Efficacy and Safety of Prophylactic Antibiotics in Preventing Ventilator-associated Pneumonia: A Randomized, Double Blind, Placebo-controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Esraa Salah Mohamed Abdallah Eladl (Other)
Responsible Party: Sponsor-Investigator, Esraa Salah Mohamed Abdallah Eladl, Assistant Lecturer of Critical Care Medicine, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD 1-11-2024
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Ventilator-Associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — beta Lactam Antibiotics

STUDY DESIGN:
Intervention Model Description: Efficacy of prophylactic antibiotic against vent.associated pneumonia
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- B.lactam (Active Comparator): Patient recieved beta lactam iv 1gm each 12h for 2 days
  Interventions: Drug: Beta Lactam Antibiotics
- Control group (Placebo Comparator): patients in the control group will receive saline iv each 12h for 2 days
  Interventions: Drug: Salin

INTERVENTIONS:
Drug: Beta Lactam Antibiotics — Beta lactam cefipim infusion (20mg/kg -12h -2 days ) total volume 10 ml
  Other Names: Cefipim
  Arms: B.lactam
Drug: Salin — Patient will receive .9 % saline (10ml /12h/2days)
  Other Names: Placebo comparator
  Arms: Control group

SUMMARY:
Evaluate efficacy and safety of prophylactic antibiotics in preventing early ventilator-associated pneumonia

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years or older

  * Both sexes will be included.
  * Invasive mechanical ventilation

Exclusion Criteria:

* ongoing pneumonia or gross aspiration confirmed by the presence of lung infiltrates on chest radiographs at admission before invasive ventilation

  * previous lung disease precluding accurate interpretation of chest radiographs
  * ongoing antibiotic therapy or during the week before admission
  * known chronic colonization with multidrug-resistant bacteria
  * known allergy to beta-lactam antibiotics
  * Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation associated pneumonia | from the 2nd to the 7th day of mechanical ventilation
  The primary outcome is the proportion of patients who will develop VAP (radiology, TLC, temperature, hemodynamic, sputum culture )from the 2nd to the 7th day of mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university hospital, Banhā, Al-Qalyubia, Egypt